CLINICAL TRIAL: NCT07284303
Title: Effect of an Automatic Infant Swing on Sleep-Wake Cycles, Comfort Behaviors, and Physiological Parameters in Newborns: A Randomized Controlled Trial
Brief Title: Infant Swing and Sleep-Wake Cycles
Acronym: AISS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Edanur Tar Bolacali, Asst. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SELCUK-2025-INFANTSWING
Record Dates: First submitted 2025-11-14; First posted 2025-12-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sleep Quality
Keywords: Bispectral Index; Comfort; Infant Swing; Newborn; Randomized Controlled Trial; Sleep-Wake Cycle
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, single-blind, two-period crossover trial conducted in a neonatal intensive care unit (NICU) in Central Anatolia, Türkiye. The study population consists of late preterm and term infants (35-42 weeks of gestation) who meet the inclusion criteria. Infants will be randomly assigned to two groups (Group A and Group B) using block randomization performed by an independent statistician. Each infant will experience both conditions - automatic swing (intervention) and standard crib (control) - in different periods according to the crossover design. The study follows the CONSORT 2010 guidelines for randomized crossover trials.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group 1: Automatic Baby Swing, Then Incubator (Experimental): The sleep, comfort, and physiological parameters of the babies in Group 1 will be assessed day and night, "First in the Automatic Baby Swing, Then in the Incubator."
  Interventions: Other: Care: Automatic Baby Swing
- Intervention Group 2: Incubator, Then in the Automatic Baby Swing (Experimental): The sleep, comfort, and physiological parameters of the babies in Group 2 will be assessed day and night, "First in the Incubator, Then in the Automatic Baby Swing."
  Interventions: Other: Care: Automatic Baby Swing

INTERVENTIONS:
Other: Care: Automatic Baby Swing — The Automatic Baby Swing aims to calm the baby by mimicking their natural movements. In this study, the low-speed "Rock-a-Bye" mode will be used because it mimics natural parental movements, making it easier for babies to fall asleep. During the implementation phase: After the baby's general condition is checked, the treatment will begin according to the group to which they were randomly assigned. If the baby is assigned to the Automatic Baby Swing, their sleep, comfort, and physiological parameters will be measured "First in the Automatic Baby Swing, Then in the Incubator" for 60 minutes during the day and night. If the baby is assigned to the other group, their sleep, comfort, and physiological parameters will be measured "First in the Incubator, Then in the Automatic Baby Swing" for 60 minutes during the day and night.

SUMMARY:
This study was planned to determine the effects of automatic baby swing application on the sleep-wake cycle, comfort behaviors and physiological parameters of babies in the neonatal intensive care unit.

DETAILED DESCRIPTION:
Sleep patterns and behavioral comfort during the neonatal period are important indicators of neurological development and physiological stability. However, noise, light, and constant medical interventions and care practices in the NICU environment can negatively affect infants' sleep continuity and quality of rest. Therefore, non-pharmacological approaches that provide sensory support, such as rhythmic and gentle rocking, are thought to be effective in promoting infant relaxation and physiological balance. In this study, an automatic baby swing with adjustable speed and rhythm will be used as an intervention to support infant comfort and sleep organization. Clinically stable term and preterm newborns who meet the specified inclusion criteria will be included in the study. Participants will be randomly assigned to two groups: the intervention group (first automatic swing application, then measurement without the swing) and the control group (first measurement without the swing, then measurement in the automatic baby swing). The intervention will be implemented for 60 minutes after daytime care at 9:00 AM and 12:00 PM, and for 60 minutes after nighttime care at 9:00 PM and 12:00 AM. The infants' BIS values, comfort, and physiological parameters will be monitored throughout the entire process. The study will evaluate the infants' sleep-wake cycles, comfort behaviors (e.g., facial expressions, body movements, crying), and physiological parameters (e.g., heart rate, respiratory rate, oxygen saturation) as outcome variables. Data will be collected using standardized observation forms and monitoring devices. This study is expected to contribute to evidence-based nursing practice by demonstrating the effects of movement-based nonpharmacological interventions on newborn comfort, sleep quality, and physiological stability.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 35-42 weeks,
* birth weight >2000-4200 grams,
* stable health status,
* spontaneous breathing,
* no sedation,
* parental volunteering to participate in the study.

Exclusion Criteria:

* - A 5-minute APGAR score below 4 at birth,
* Requirement of resuscitation,
* Presence of a congenital anomaly,
* Requirement of interventional intervention in the head region,
* Presence of central nervous system dysfunction,
* Presence of postpartum medical complications.

Exclusion Criteria (during the research):

Sudden need for resuscitation Sudden deterioration of the stabilization of health status

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1: COMFORTneo Total Score | At 0, 30, and 60 minutes.
  The COMFORTneo scale assesses seven behavioral and physiological parameters (muscle tone, alertness, facial tension, calmness/agitation, body movements, respiratory response, and crying). These parameters will be combined to produce a single total score (range 6-30). Only the total score will be reported.

SECONDARY OUTCOMES:
Secondary Outcome 1: Infant Body Temperature | At 0, 30, and 60 minutes.
  Infant axillary body temperature measured in degrees Celsius (°C).
Secondary Outcome 2: Infant Heart Rate | At 0, 30, and 60 minutes.
  Infant heart rate measured in beats per minute.
Secondary Outcome 3: Infant Respiratory Rate | At 0, 30, and 60 minutes.
  Infant respiratory rate measured in breaths per minute.
Secondary Outcome 4: Infant Oxygen Saturation | At 0, 30, and 60 minutes.
  Pulse oximetry oxygen saturation measured as %SpO₂.
Secondary Outcome 5: Infant Blood Pressure | At 0, 30, and 60 minutes.
  Non-invasive systolic and diastolic blood pressure measured in mmHg.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yasova Barbeau D, Krueger C, Huene M, Copenhaver N, Bennett J, Weaver M, Weiss MD. Heart rate variability and inflammatory markers in neonates with hypoxic-ischemic encephalopathy. Physiol Rep. 2019 Aug;7(15):e14110. doi: 10.14814/phy2.14110. PMID 31397094
- [Result] van Dijk M, Roofthooft DW, Anand KJ, Guldemond F, de Graaf J, Simons S, de Jager Y, van Goudoever JB, Tibboel D. Taking up the challenge of measuring prolonged pain in (premature) neonates: the COMFORTneo scale seems promising. Clin J Pain. 2009 Sep;25(7):607-16. doi: 10.1097/AJP.0b013e3181a5b52a. PMID 19692803
- [Result] Huang Q, Lai X, Liao J, Tan Y. Effect of non-pharmacological interventions on sleep in preterm infants in the neonatal intensive care unit: A protocol for systematic review and network meta-analysis. Medicine (Baltimore). 2021 Oct 29;100(43):e27587. doi: 10.1097/MD.0000000000027587. PMID 34713833
- [Result] Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. BMJ. 2019 Jul 31;366:l4378. doi: 10.1136/bmj.l4378. PMID 31366597
- [Result] Caba-Flores MD, Ramos-Ligonio A, Camacho-Morales A, Martinez-Valenzuela C, Viveros-Contreras R, Caba M. Breast Milk and the Importance of Chrononutrition. Front Nutr. 2022 May 12;9:867507. doi: 10.3389/fnut.2022.867507. eCollection 2022. PMID 35634367